CLINICAL TRIAL: NCT04243317
Title: A Pilot Study to Assess the Feasibility and Adherence of a Sleep Improvement Intervention for Weight Loss and Its Maintenance in Sleep Impaired Obese Adults
Brief Title: Feasibility of a Sleep Improvement Intervention for Weight Loss and Its Maintenance in Sleep Impaired Obese Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zayed University (Other)
Collaborators: Al Jalila Children's Specialty Hospital (Other); Imperial College London Diabetes Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZU18_102_F
Record Dates: First submitted 2019-12-02; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Obesity
Keywords: sleep
MeSH Terms: conditions — Obesity | interventions — Diet; Sleep

STUDY DESIGN:
Intervention Model Description: Those with sleep impairment (sleep duration of ≤6.5hours per 24-hours; and/or poor sleep quality [<85% efficiency]; and/or misaligned nocturnal sleep timing [>03:00 on weekdays]) who are also obese (BMI ≥27.5 kg/m2) will be recruited and randomized to a 12-week weight loss intervention with/without sleep improvement. Volunteers will be followed for a further six months to assess multiple outcome measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The control group will adhere to a 1200 kcal restriction daily for 12 weeks.
  Interventions: Behavioral: Lifestyle & diet
- Experimental (Experimental): The experimental group will adhere to a 1200 kcal restriction daily for 12 weeks and will maintain sleep improvement
  Interventions: Behavioral: Lifestyle, diet & sleep

INTERVENTIONS:
Behavioral: Lifestyle & diet — The control group will receive lifestyle and dietary advice accompanied by meal replacements and dietary plans.
  Arms: Control
Behavioral: Lifestyle, diet & sleep — The control group will receive lifestyle and dietary advice accompanied by meal replacements and dietary plans. The experimental group will additionally receive a sleep improvement program based on CBTi.
  Arms: Experimental

SUMMARY:
The primary objective of the proposed study is to develop, deliver and assess the feasibility and adherence to a targeted behavioral sleep intervention for sleep impaired obese patients.

Secondary objectives are to demonstrate that a targeted behavioral sleep intervention can improve treatment outcomes in obese adult outpatients enrolled to a lifestyle and dietary modification program; and to demonstrate that a targeted behavioral sleep intervention enhances the long-term maintenance of treatment gains in obese adults enrolled in a lifestyle and dietary modification program.

Those with sleep impairment (sleep duration of ≤6.5hours per 24-hours; and/or poor sleep quality [<85% efficiency]; and/or misaligned nocturnal sleep timing [>03:00 on weekdays]) who are also obese (Body Mass Index [BMI] ≥27.5 kg/m2) will be recruited and randomized to a 12-week weight loss intervention with/without sleep improvement. Volunteers will be followed for a further six months to assess multiple outcome measures.

It is hypothesised that inclusion of a targeted behavioral sleep improvement intervention will be feasible and acceptable and will enhance immediate and long-term treatment outcomes of obese adults enrolled to a lifestyle and dietary modification program. The results of the study will be used to better inform the design and development of a future Randomized Controlled Trial (RCT).

Sleep improvement may be incorporated into weight management treatments as a cost-effective alternative/addition.

DETAILED DESCRIPTION:
The primary objective of the proposed study is to develop, deliver and assess the feasibility and adherence to a targeted behavioral sleep intervention for sleep impaired obese patients.

Secondary objectives are to demonstrate that a targeted behavioral sleep intervention can improve treatment outcomes in obese adult outpatients enrolled to a lifestyle and dietary modification program; and to demonstrate that a targeted behavioral sleep intervention enhances the long-term maintenance of treatment gains in obese adults enrolled in a lifestyle and dietary modification program.

Those with sleep impairment (sleep duration of ≤6.5hours per 24-hours; and/or poor sleep quality [<85% efficiency]; and/or misaligned nocturnal sleep timing [>03:00 on weekdays]) who are also obese (Body Mass Index [BMI] ≥27.5 kg/m2) will be recruited and randomized to a 12-week weight loss intervention (based on a previously developed specialist lifestyle management program) with/without sleep improvement (based on a cognitive behaviour treatment developed to treatment sleep problems in US military). Volunteers will be followed for a further six months to assess multiple outcome measures. Other secondary measures to be assessed are mood (Hospital Anxiety Depression Scale [HADS], food intake (24-hour food recall), quality of life (IWQOL-LITE & EQ-5D), and sleep (PSQI & RU_SATED), all of which will be assessed using validated questionnaires that have been previously assessed for reliability.

It is hypothesised that inclusion of a targeted behavioral sleep improvement intervention will be feasible and acceptable and will enhance immediate and long-term treatment outcomes of obese adults enrolled to a lifestyle and dietary modification program. The results of the study will be used to better inform the design and development of a future Randomized Controlled Trial (RCT).

Sleep improvement may be incorporated into weight management treatments as a cost-effective alternative/addition.

ELIGIBILITY:
Inclusion Criteria:

* Sleep impaired individuals defined as meeting one or more of the following objectively estimated sleep feature: 1) ≤6.5hours per 24-hours; 2) poor sleep quality (<85% efficiency); 3) misaligned nocturnal sleep timing (>03:00 on weekdays);
* Obese (BMI ≥27.5 kg/m2 for Asians/Arabs or BMI ≥30.0 kg/m2 for Europeans/Caucasians);
* Men/women;
* Age 18-50 years (upper age limit chosen due to specific alterations in sleep duration and quality commonly observed after this age);
* Good English language comprehension/communication skills;
* Able to provide informed consent and willing to participate in the study.

Exclusion Criteria:

* Currently taking medication(s) that may interfere with weight loss (e.g. corticosteroids);
* Contraindications to use of the Cambridge Weight Plan (heart attack or stroke three months preceding study participation; lactose intolerance; gallstones; porphyria; active gout);
* Medications that may interfere with sleep;
* Clinically diagnosed sleep disorder(s) or those at high risk of undiagnosed OSA based on three questionnaires (Berlin, ESS, STOP-BANG);
* Chronic illness (asthma, COPD, diabetes, arthritis, fibromyalgia, heart condition, kidney or liver disease);
* Uncontrolled hypertension;
* Polycystic ovary syndrome;
* Endocrine disorder(s), except for stable treated hypothyroidism;
* Psychiatric disorder(s), except for stable treated depression;
* Currently taking monoamine oxidase inhibitor medication;
* Previous/planned bariatric surgery;
* Diagnosed eating disorders;
* Night-shift workers;
* Substance use;
* Excessive alcohol consumption;
* Known pregnancy or planned pregnancy during the study/breastfeeding or given birth in last 3 months;
* Family circumstances e.g. infants, young children, pets that will make study adherence difficult.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Body weight (kg) | 3 months
  Amount of group weight loss by group will be calculated and compared at the end of the 12-week intervention period

SECONDARY OUTCOMES:
Hospital Anxiety & Depression Scale (HADS) | 6 months
  Mood will be assessed using the HADS and changes in scores will be compared (baseline v post-intervention) at an individual and group level. Higher scores indicate higher levels of abnormality and the score range is 0-21, with defined cut points where 0-7=normal, 8-10=borderline and 11-21=abnormal for both anxiety and depression
Body weight (kg) loss maintenance | 6 months
  It will be assessed which group maintains weight loss at the 6-month follow-up, post the 12-week intervention
Impact of Weight on Quality of Life (IWQOL-LITE) | 6 months
  The IWQOL-LITE is a 31-item self-reported weight-related quality of life measure covering 5 domains. Changes in the total score and each of the scores on the five domains on the IWQOL-LITE will be examined at an individual and group level and comparisons will be made across the two groups in the study. The range of scores are 0-100 with lower scores indicating greater impairment

CONTACTS AND LOCATIONS:
Locations (1):
- Zayed University, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
IPD will only be shared with researchers within the same research team who are listed on the approval ethics application
Supporting Information: Study Protocol, CSR
Time Frame: This information will be shared with other members of the research team who are approved on the ethics application. The information will be available to the research team throughout the course of the study.
Access Criteria: The master file will be retained by the PI and stored on a password-protected computer. Access will only be permitted to other members of the research team for study related activities.

DOCUMENTS (1):
  • Informed Consent Form (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT04243317/ICF_000.pdf